CLINICAL TRIAL: NCT06727955
Title: Prospective Cohort Study on Predicting the Progression of Diabetic Microangiopathy Using Multimodal Eye Imaging
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2023514
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; artificial intelligence model; multimodal eye imaging
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To develop an artificial intelligence (AI) model to predict DR progression based on a prospective cohort database.With use of an innovative AI model and a validated machine learning algorithm, based on multimodal vascular and neuro imaging of the eye, the progression of diabetic microangiopathy especially the DR could successfully be predictse and fundamentally facilitate diabetes management.

DETAILED DESCRIPTION:
To develop an artificial intelligence (AI) model to predict DR progression based on a prospective cohort database.This study will first conduct a prospective single-center cohort, which will enroll 250 type 2 diabetes mellitus patients with non-proliferative diabetic retinopathy (NPDR). The follow-up time points will be 3 months, 6 months, 1 year, 2 years, and 3 years after enrollment or reaching the endpoint (any condition that needs retinal photocoagulation, anti-vascular endothelial growth factor injections, and pars plana vitrectomy). The study will collect both patient clinical characteristics and multi-model eye imaging. With use of an innovative AI model and a validated machine learning algorithm, based on multimodal vascular and neuro imaging of the eye, the progression of diabetic microangiopathy especially the DR could successfully be predictse and fundamentally facilitate diabetes management.

ELIGIBILITY:
Inclusion Criteria:

* (1) age between 40 and 80 years, regardless of gender, (2) meet the diagnostic criteria of T2DM based on the Standards of Medical Care in Diabetes (2021)11, and complete evaluation at the Endocrinology Department of Peking University Third Hospital, (3) meet the Diabetic Retinopathy Severity Scale (DRSS) score level of mild to moderate-severe NPDR (i.e. 35 ≤ DRSS level ≤ 60, as shown in eTables 1 & 2 in the Supplement) based on the montages ultra-widefield (UWF) fundus photographs,12 without clinically significant macular edema (CSME, defined as one or more of the followings: retinal thickening at or within 500 μm of the center of the macula; hard exudates at or within 500 μm of the center of the macula, if associated with adjacent retinal thickening; or a zone or zones of retinal thickening one disc area in size, at least part of which is within one disc diameter of the center of the macula),13 (4) willing to sign the informed consent form.

Exclusion Criteria:

* (1) conjunctivitis, keratitis, blepharitis, episcleritis, scleritis, uveitis, severe dry eye disease, using anti-glaucoma eyedrops, or any condition causing conjunctival congestion or ciliary congestion, (2) pterygium, wearing contact lens in the past week, ocular surface burn, conjunctival tumors, or any condition causing significant conjunctival vascular deformities, (3) previously undergone intraocular surgeries involving manipulation of the conjunctiva, or corneal refractive surgery, (4) history of hematological disorder, dysthyroidism, rheumatic disorder, malignant tumor, (5) refractive media opacity resulting in poor visualization of fundus photographs, (6) difficulty in maintaining fixation or comprehension, making it challenging to cooperate with the examination, (7) difficulty in completing follow-up visits in 3 years.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. age between 40 and 80 years, regardless of gender,
  2. meet the diagnostic criteria of T2DM based on the Standards of Medical Care in Diabetes (2021)11, and complete evaluation at the Endocrinology Department of Peking University Third Hospital,
  3. meet the Diabetic Retinopathy Severity Scale (DRSS) score level of mild to moderate-severe NPDR (i.e. 35 ≤ DRSS level ≤ 60, as shown in eTables 1 & 2 in the Supplement) based on the montages ultra-widefield (UWF) fundus photographs,12 without clinically significant macular edema (CSME, defined as one or more of the followings: retinal thickening at or within 500 μm of the center of the macula; hard exudates at or within 500 μm of the center of the macula, if associated with adjacent retinal thickening; or a zone or zones of retinal thickening one disc area in size, at least part of which is within one disc diameter of the center of the macula),13
  4. willing to sign the informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
DRSS Score and Classification | At Enrollment
  The progression of DR is based on the increase of DRSS score and classification.
  Ophthalmologists at the Department of Ophthalmology, Peking University Third Hospital, will independently read UWF CFP in a semi-quantitative manner to assess the severity of DR based on the DRSS.
  Progression of DR in T2DM patients with varying degrees of NPDR is calculated based on DRSS. An increase of at least one level in grading is considered progression. For instance, progression from grade 43A to 47A or higher is considered progression, while progression from 43A to 43B is not.

SECONDARY OUTCOMES:
Renal Function Test | At Enrollment
  Progression to DN is considered when the UACR increases from < 30 mg/g to ≥ 30 mg/g.
Peripheral Neuropathy Assessment | At Enrollment
  Progression to DPN is considered when the MNSI score questionnaire section ≥ 4 points, while the examination section ≥ 2 points.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Qi, Dr., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China